CLINICAL TRIAL: NCT01324518
Title: Safety and Efficacy of ORM-12741 on Cognitive and Behavioral Symptoms in Patients With Alzheimer's Disease
Brief Title: Safety and Efficacy of ORM-12741 in Patients With Alzheimer's Disease
Acronym: ALPO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3098006
Record Dates: First submitted 2011-03-24; First posted 2011-03-29 (Estimated); Results first posted 2021-04-28 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — ORM-12741

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low dose of ORM-12741 (Experimental)
  Interventions: Drug: ORM-12741
- High dose of ORM-12741 (Experimental)
  Interventions: Drug: ORM-12741
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo for ORM-12741

INTERVENTIONS:
Drug: ORM-12741 — 60mg twice a day
  Arms: Low dose of ORM-12741
Drug: ORM-12741 — 200mg twice a day
  Arms: High dose of ORM-12741
Drug: Placebo for ORM-12741 — Placebo twice a day
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether ORM-12741 is safe and effective in the treatment of Alzheimer's disease.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether ORM-12741 is safe and effective in the treatment of cognitive and behavioral symptoms in patients with Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained from the patient and legally acceptable representative, if required
* Informed consent obtained from the caregiver
* Males and and females between 55-90 years
* Diagnosis of probable Alzheimer's disease, history of progressive cognitive deterioration
* Brain imaging consistent with Alzheimer's disease
* Mini-mental state examination score 12-21
* Treated with donepezil, rivastigmine or galantamine
* At least mild level of behavioral symptoms

Exclusion Criteria:

* Other types of dementias
* Modified Hachinski Ischemia Score > 4
* Use of memantine, antipsychotics, anticholinergic medication and benzodiazepines (at a max of 3 nights/week) within 2 months
* Changes in antidepressant dosing within 2 months
* Use of other psychotropic agents
* Myocardial infarction within the past 2 years
* Malignancy within the past 5 years
* Suicidal ideation, risk of suicide
* History of alcoholism or drug abuse within 5 years
* Clinically significant cardiovascular, pulmonary, gastrointestinal, hepatic, renal, neurological or psychiatric disorder or any other major concurrent illness
* Specific findings in brain imaging
* Abnormal findings in heart rate, blood pressure, ECG, laboratory tests, physical examination; orthostatic hypotension
* Blood donation or participation in a drug study within 60 days
* Previous AD immunotherapy treatment
* Patient cannot complete the computerised cognitive training
* Patients who reside in a skilled nursing facility
* Patients who are not able to swallow capsules

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2012-09 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juha Rinne, Prof, Principal Investigator — Clinical Research services Turku (CRST)
Locations (1):
- Clinical Research Services Turku (CRST), Turku, Finland

REFERENCES:
- See also: AAN 65th ANNUAL MEETING ABSTRACT — https://www.aan.com/PressRoom/Home/GetDigitalAsset/10708

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 4 countries (18 centres): Finland, Poland, Romania and Spain. Of these, 1 centre screened but did not randomise any subjects. Study period was 27 Apr 2011-21 Sep 2012 (first subject first visit to last subject last visit).
Pre-assignment Details: A total of 132 subjects were screened and 100 were randomized to 3 treatment groups. 30 patients were excluded prior randomization due to inclusion/exclusion criteria, 2 due to personal reasons.
Period: Overall Study
Arm/Group | Low Dose of ORM-12741 | High Dose of ORM-12741 | Placebo
Started | 33 | 33 | 34
Completed | 28 | 30 | 33
Not Completed | 5 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose of ORM-12741 | High Dose of ORM-12741 | Placebo | Total
Number analyzed (Participants) | 33 | 33 | 34 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.8 (8.2) | 71.8 (6.8) | 72.3 (8.5) | 72.0 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 23 | 17 | 59
  Male | 14 | 10 | 17 | 41

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Adverse events from start of ORM-12741 treatment until end of study visit.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose of ORM-12741 | High Dose of ORM-12741 | Placebo
Number analyzed (Participants) | 33 | 33 | 34
Participants | 18 | 21 | 21

2. Primary Outcome: Quality of Episodic Memory
Description: The Cognitive Drug Research (CDR) computerised battery tests is designed to evaluate the effects of novel compounds on the quality of cognitive functioning. Quality of Episodic Memory measures the capability of maintaining information in episodic memory and is assessed as the sum of sensitivity indices from 4 memory tasks on the CDR computerised battery tests. Values are calculated by a computer and higher scores mean better outcome.
Time Frame: 3 months
Population: per protocol population
Measure: Mean (Standard Deviation); unit: Index score
Arm/Group | Low Dose of ORM-12741 | High Dose of ORM-12741 | Placebo
Number analyzed (Participants) | 24 | 26 | 28
Index score | 100.7 (92.2) | 85.0 (59.6) | 46.3 (62.4)

3. Primary Outcome: Quality of Working Memory
Description: The Cognitive Drug Research (CDR) computerised battery tests is designed to evaluate the effects of novel compounds on the quality of cognitive functioning. Quality of Working Memory measures the capability of maintaining information in working memory and is assessed as the sum of sensitivity indices from 2 memory tasks on the CDR computerised battery tests. Values are calculated by a computer and higher scores mean better outcome.
Time Frame: 3 months
Population: per protocol population
Measure: Mean (Standard Deviation); unit: Index score
Arm/Group | Low Dose of ORM-12741 | High Dose of ORM-12741 | Placebo
Number analyzed (Participants) | 24 | 26 | 28
Index score | 1.20 (0.53) | 1.18 (0.47) | 0.82 (0.59)

4. Primary Outcome: Quality of Memory
Description: The Cognitive Drug Research (CDR) computerised battery tests is designed to evaluate the effects of novel compounds on the quality of cognitive functioning. Quality of Memory is a combination of outcome measures Quality of Working Memory & Quality of Episodic Memory. Values are calculated by a computer and higher scores mean better outcome.
Time Frame: 3 months
Population: per protocol population
Measure: Mean (Standard Deviation); unit: Index score
Arm/Group | Low Dose of ORM-12741 | High Dose of ORM-12741 | Placebo
Number analyzed (Participants) | 24 | 26 | 28
Index score | 216.53 (133.15) | 196.37 (93.72) | 117.15 (104.30)

5. Primary Outcome: Speed of Memory
Description: The Cognitive Drug Research (CDR) computerised battery tests is designed to evaluate the effects of novel compounds on the quality of cognitive functioning. Speed of Memory is assessed as the sum of speed measures from 2 memory tasks and 2 recognition tasks on the CDR computerised battery tests. Values are calculated by a computer and higher scores mean better outcome.
Time Frame: 3 months
Population: per protocol population
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Low Dose of ORM-12741 | High Dose of ORM-12741 | Placebo
Number analyzed (Participants) | 24 | 26 | 28
msec | 8287.8 (3898.2) | 8930.30 (5379.5) | 8082.2 (4064.1)

6. Primary Outcome: Power of Attention
Description: The Cognitive Drug Research (CDR) computerised battery tests is designed to evaluate the effects of novel compounds on the quality of cognitive functioning. Power of attention measures speed and attention and is assessed from 3 attentional tasks on the CDR computerised battery tests. Values are calculated by a computer and higher scores mean better outcome.
Time Frame: 3 months
Population: per protocol population
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Low Dose of ORM-12741 | High Dose of ORM-12741 | Placebo
Number analyzed (Participants) | 25 | 26 | 28
msec | 1940.3 (533.3) | 1978.0 (1040.4) | 2077.9 (995.8)

7. Primary Outcome: Continuity of Attention
Description: The Cognitive Drug Research (CDR) computerised battery tests is designed to evaluate the effects of novel compounds on the quality of cognitive functioning. Continuity of attention measures speed and accuracy and is calculated from 3 attentional tasks on the CDR computerised battery tests. Values are calculated by a computer and higher scores mean better outcome.
Time Frame: 3 months
Population: per protocol population
Measure: Mean (Standard Deviation); unit: Index score
Arm/Group | Low Dose of ORM-12741 | High Dose of ORM-12741 | Placebo
Number analyzed (Participants) | 25 | 26 | 28
Index score | 85.7 (11.0) | 84.8 (15.3) | 79.7 (21.2)

8. Secondary Outcome: NPI Total Score
Description: The total score of Neuropsychiatric Inventory (NPI) was assessed by a caregiver interview. 10 behavioral areas were included: Delusions, Hallucinations, Agitation/Aggression, Depression/Dysphoria, Anxiety, Elation/Euphoria, Apathy/Indifference, Disinhibition, Irritability/Lability, and Aberrant Motor Behaviour. Higher scores mean worse outcome. Minimum value 0, maximum value 120.
Time Frame: 3 months
Population: per protocol population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low Dose of ORM-12741 | High Dose of ORM-12741 | Placebo
Number analyzed (Participants) | 25 | 26 | 28
score on a scale | 14.7 (9.1) | 13.7 (8.9) | 20.2 (19.0)

9. Secondary Outcome: Caregiver Distress Score
Description: Caregiver distress score generated by adding together the scores of individual NPI distress questions of Neuropsychiatric Inventory NPI. Higher scores mean worse outcome. Minimum value 0, maximum value 120.
Time Frame: 3 months
Population: per protocol population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low Dose of ORM-12741 | High Dose of ORM-12741 | Placebo
Number analyzed (Participants) | 25 | 26 | 28
score on a scale | 9.2 (6.0) | 8.0 (4.3) | 11.0 (10.4)

10. Secondary Outcome: Pharmacokinetics of ORM-12741
Description: ORM-12741 plasma trough concentrations at week 12.
Time Frame: 3 months
Population: M-ITT population
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Low Dose of ORM-12741 | High Dose of ORM-12741 | Placebo
Number analyzed (Participants) | 29 | 31 | 32
ng/ml | 18.4 (13.9) | 61.0 (45.9) | 0 (0)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Low Dose of ORM-12741 | High Dose of ORM-12741 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/33 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/33 | 1/33 | 0/34
Other Adverse Events (participants affected / at risk) | 8/33 | 14/33 | 16/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose of ORM-12741 (N=33) | High Dose of ORM-12741 (N=33) | Placebo (N=34)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) — Cholestatic syndrome
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose of ORM-12741 (N=33) | High Dose of ORM-12741 (N=33) | Placebo (N=34)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 1 (1) | 2 (3)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 3 (5)
Vomiting (Gastrointestinal disorders) | 1 (1) | 4 (6) | 1 (1)
Irritability (General disorders) | 0 (0) | 2 (2) | 3 (3)
Urinary tract infection (Infections and infestations) | 1 (2) | 5 (5) | 3 (3)
Headache (Nervous system disorders) | 2 (4) | 1 (1) | 4 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No